CLINICAL TRIAL: NCT00592826
Title: Phase III Study of the Usability of the HMP Device
Brief Title: HMP (Home Macular Perimeter) -Usability Trial
Status: Completed | Type: Observational
Sponsor: Notal Vision Ltd. (Industry)
Responsible Party: Sponsor
Organization: Notal Vision Inc. (Industry)
Other Study IDs: T3; WIRB Pr. No.: 20071980
Record Dates: First submitted 2008-01-01; First posted 2008-01-14 (Estimated); Last update posted 2015-04-14 (Estimated); Status verified 2015-04

CONDITIONS: Age Related Macular Degeneration
Keywords: PHP; HMP; HPHP; AMD; CNV
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The study is divided in two stages. The purpose of the first stage is to evaluate the percentage of subjects that can unpack the device, install it, learn the task and calibrate it according to their personal capabilities. The purpose of the second stage is to assess the ability of the subjects to perform reliable tests .

DETAILED DESCRIPTION:
Stage I:

* Receive a packed HMP device.
* Unpack the device and install it, using a set-up guide
* Use an interactive tutorial to learn the task
* Calibrate the sensitivity of the test

This stage will be completed within 1 to 5 visits, depending on personal progress rate.

Subjects who have successfully completed stage I will be recruited to stage II.

Those subjects will:

• Perform 3 tests , each test in a different day

ELIGIBILITY:
Inclusion Criteria:

* Age >50 years
* Familiar with computer usage
* Capable and willing to sign a consent form and participate in the study
* Ability to speak, read and understand instructions in English

Exclusion Criteria:

* Subject already participating in another study.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects will be recruited in community centers and clinics and will include up to 25 people aged >50 years (Age-related Macular Degeneration age group). The group will be heterogeneous in terms of education, age, ethnic background, and gender. The subjects will be enrolled in one site in the USA In order to get 20 completed subjects, and based of assumption of 25% attrition- 25 subjects will be recruited to the study
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2007-11; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects who successfully set up the device | 1 month
Proportion of subjects who successfully pass the training program (successful calibration module) | 1 month

SECONDARY OUTCOMES:
Proportion of subjects with reliable tests results | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Adam Mr Weinstein, MD, Principal Investigator — Kidney Health Center of Maryland